CLINICAL TRIAL: NCT01209507
Title: A Prevalence Study of Adrenal Suppression After Adjuvant Corticosteroid Administration During Gynecologic Cancer Chemotherapy
Brief Title: Prevalence Study of Adrenal Suppression After Corticosteroids During Chemotherapy
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 10-0190.cc
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Adrenal Suppression
Keywords: Adrenal suppression; Chemotherapy fatigue; Quality of life
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chemotherapy every 3 weeks: One treatment of chemotherapy every 3 weeks. Chemotherapy will either be 2 doses of 20 mg orally (PO) (12 hrs prior and immediately before treatment) or 1 dose via IV. The total dose per cycle is 20-40 mg every 3 weeks for 18 weeks.
  Interventions: Other: Chemotherapy
- Weekly chemotherapy: Chemotherapy will be given three times in a three week cycle. Chemotherapy will be given either Day 1, 8, and day 15 or Day 1,2 and day 8). Chemotherapy will either be 2 doses of 20 mg PO (12 hrs priors and immediately before treatment) or 1 dose via IV. The total dose per cycle will be 20-40 mg approximately for 18 weeks.
  Interventions: Other: Chemotherapy

INTERVENTIONS:
Other: Chemotherapy — This study is designed only to look at the prevalence of adrenal suppression during chemotherapy. If adrenal suppression is detected, treatment will be off-study at the treating physician's discretion.
  Other Names: Adrenal Suppression

SUMMARY:
Gynecologic Oncology patients have several different chemotherapy regimens, and dexamethasone is now routinely given to prevent allergic reactions to the chemotherapeutic agents. The most common chemotherapeutic agents used are paclitaxel and carboplatin. This combination regimen is given every three weeks for a total of 5-6 doses. Each dose is given after administration of 20 mg dexamethasone twelve hours prior to and the morning of chemotherapy. Dexamethasone is used for its antiemetic effects, but also to minimize the potentially fatal hypersensitivity reaction that can occur with paclitaxel. Another commonly used chemotherapy regimens is weekly cisplatin given with one dose of dexamethasone for cervical cancer. Chronic steroids are known to cause adrenal suppression, but it is not known if the amount of dexamethasone given with the gynecologic cancer chemotherapy regimens described above causes adrenal insufficiency in these patients. The investigators hypothesis is that some women receiving steroids with their chemotherapy may have adrenal insufficiency, and that they will have greater than normal chemotherapy-related fatigue.

DETAILED DESCRIPTION:
This is a non-blinded, non-randomized, non-interventional prospective cohort study to evaluate the prevalence of adrenal suppression in gynecologic cancer patients undergoing chemotherapy regimens requiring concurrent dexamethasone. Women with gynecologic cancers (including cervical, endometrial, ovarian, fallopian tube, or primary peritoneal cancers) who are scheduled to begin chemotherapy with any of the standard chemotherapy regimens that also receive dexamethasone. After informed consent is obtained, they will have peripheral blood samples drawn at the time of routine blood draw for (ideally a fasting morning) cortisol level at three different times in their routine care. Patients will also answer a quality of life questionnaire at the times of these blood draws to assess for symptoms associated with treatment (nausea, vomiting, fatigue). A total of 80 subjects will be recruited to participate. 40 subjects will be given chemotherapy regimens receiving dexamethasone with three chemotherapy treatments in a three week cycle. 40 subjects will be given chemotherapy regimens receiving dexamethasone with one chemotherapy treatment in a three week cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have age greater or equal to 18
2. Patients with histologic diagnosis of cervical, endometrial, or ovarian cancer who are receiving chemotherapy
3. Any clinical stage allowed
4. GOG performance status 0, 1, or 2
5. Written informed consent and HIPAA authorization obtained prior to any initiation of study procedures

Exclusion Criteria:

1. The presence of other comorbid conditions known to impact adrenal function, whether primary adrenal dysfunction, or dysfunction due to administration of steroids for treatment (Addison's or Cushings disease, pituitary or hypothalamic disease, systemic lupus erythematosis, rheumatoid arthritis, asthma)
2. Patients who have received chronic or pulsed steroids within the past 9 months.
3. Patients with previous diagnosis of adrenal suppression.
4. Underlying psychiatric condition which would, in the opinion of the investigator, preclude compliance with study requirements
5. Women who are pregnant are not eligible to participate.
6. Patients who have received prior radiotherapy or chemotherapy for an abdominal or pelvic tumor are excluded. Prior radiation or adjuvant chemotherapy for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than 3 years prior to registration, and the patient remains free of recurrent or metastatic disease.
7. Patients with invasive malignancies, with exception of non-melanoma skin cancer, and specific malignancies noted above, who had (or have) any evidence of other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be open to all women over the age of 18 scheduled to begin standard of care chemotherapy for a gynecologic malignancy, either every 3 weeks (carboplatin and taxol) or weekly (cisplatin). The study is restricted by gender due to the population of interest being women with gynecologic malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Identify the level of adrenal suppression with recurrent, intermittent steroid administration during gynecologic chemotherapy regimens in all participating patients | 6 months
  This will be done by testing a morning cortisol level in patients at the time of routine blood draw at three different time points in each patient's chemotherapy regimen.

SECONDARY OUTCOMES:
Identify the differences in quality of life scores among patients with adrenal suppression and those with normal function | 6 months
  Differences in quality of life scores will be measured using a modified FACT-G questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Monique A Spillman, MD, Principal Investigator — University of Colorado Denver Anschutz Medical Center
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No